CLINICAL TRIAL: NCT05275218
Title: Effect of an Extended "Kidney Disease: Improving Global Outcomes" (KDIGO) Bundle Versus Standard of Care Therapy on Persistent Acute Kidney Injury in High-risk Patients After Major Surgery
Brief Title: Effect of an Intervention to Prevent Acute Kidney Injury Versus Standard Care in High-risk Patients After Major Surgery
Acronym: PrevProgAKI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08-AnIt-21
Record Dates: First submitted 2022-02-17; First posted 2022-03-11 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Acute Kidney Injury (Nontraumatic)
Keywords: surgery; biomarker; CCL14 protein
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Implementation of the KDIGO bundle for at least 72 hours 1. Discontinuation of all nephrotoxic drugs when possible 2. Optimization of volume status and perfusion pressure. 3. Consideration of a functional hemodynamic monitoring. 4.Close monitoring of serum creatinine, and urinary output 5. Avoidance of hyperglycemia 6. Considerations of alternatives to radiocontrast agents 7. Non-invasive or invasive diagnostic workup 8. Nephrology consultation.
  Interventions: Procedure: Implementation of the KDIGO bundle)
- Control Group (No Intervention): Patients in the control group will receive standard of care. According to best clinical practice, this includes the following targets (unless specific individual targets are chosen by treating physician):
  * mean arterial pressure (MAP): ≥ 65 mmHg
  * passive leg raising test (PLRT): increase of cardiac output (CO)<10%

INTERVENTIONS:
Procedure: Implementation of the KDIGO bundle) — Comprehensive Implementation of the Bundle recommended by the "Kidney Disease: Improving Global Outcomes Group "(KDIGO bundle)
  Arms: Intervention Group

SUMMARY:
There is no specific therapy for acute kidney injury. It is presumed that supportive measures improve the care and outcome of patients with acute kidney injury.

To investigate whether an implementation of a supportive extended care "bundle" in high-risk patients for persistent acute kidney injury (AKI) can reduce the occurrence of persistent surgical AKI.

In order to investigate whether the extended KDIGO bundle can prevent persistent AKI in patients with high chemokine ligand 14 (CCL14) as well as in patients with low CCL14, patients will be randomized with stratification by the CCL-value.

DETAILED DESCRIPTION:
All patients will receive standard of care therapy according to the standards of our center. After identifying surgical patients with a moderate or severe (stage 2 or 3) AKI patients will be randomly allocated to the control or intervention group according to the CCL14 results which will be measured as part of the study. According to the literature, patients with a CCL14 <1.3ng/ml are at low risk of progression and patients with a CCL14≥1.3ng/ml are at high risk of AKI progression. In order to have both patient groups included, we will have two groups (patients at low and at high risk of AKI progression) and these will be randomized to receive either standard of care or an extended KDIGO bundle (in total 4 groups).

Control intervention / reference test: Patients in the control groups will be treated according to the standard of care. The only two hemodynamic targets in this group are the mean arterial pressure (mean arterial pressure (MAP)>65mmHg) and passive leg raising test (PLRT) (increase of cardiac output (CO) <10%).

In the intervention groups, an extended KDIGO guideline bundle will be implemented (Discontinuation of all nephrotoxic agents when possible, optimization of volume status and perfusion pressure, consideration of a functional hemodynamic monitoring, close monitoring of serum creatinine and urine output, avoidance of hyperglycemia, consideration of alternatives to radio contrast agents, non-invasive or invasive diagnostic workup, nephrology consultation)

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥18 years)
2. Moderate or severe AKI ((defined by the 2012 KDIGO criteria, KDIGO stage 2 and 3), determined by either serum creatinine or urine output) within 72h after a surgical procedure
3. Written informed consent

Exclusion Criteria:

1. Dialysis-dependent chronic kidney disease
2. Prior kidney transplant
3. Infections with human immunodeficiency virus or hepatitis
4. Hepatorenal syndrome
5. Pregnancy or breast-feeding
6. Participation in another interventional trial that investigates a drug that affects the kidney function within the last 3 months
7. Persons held in an institution by legal or official order
8. Persons with any kind of dependency on the investigator or employed by the responsible institution or investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of persistent severe AKI | 72 hours after start of intervention
  The primary endpoint is the development of persistent severe (stage 3) AKI lasting for at least 72h defined as ≥3-fold increase in serum creatinine in relation to baseline or serum creatinine ≥4.0mg/dl with an acute increase of 0.5mg/dl or a decrease in urine output <0.3ml/kg/h for 24 hours or anuria for 12 hours. Persistent AKI is defined as follows: patients with stage 3 AKI at enrollment require a persistence of 72h or more to meet the endpoint. Patients enrolled at stage 2 AKI require a progression to stage 3 within 48 hours and a persistence at stage 3 for 72 consecutive hours to be considered endpoint positive. Additionally, patients with severe AKI who fail to achieve 72h due to death or the initiation of renal replacement therapy are considered endpoint positive as well

SECONDARY OUTCOMES:
Number of patients with major adverse kidney events (MAKE) | 90 days after start of intervention
  Composite endpoint consisting of death or initiation of renal replacement therapy within 90 days or persistent renal dysfunction (defined as a decrease in estimated glomerular filtration rate (eGFR) to < 75% of baseline)
  - The baseline serum creatinine is taken as the value obtained prior to the day of operation
Length of intensive care unit stay | up to 90 days after start of intervention
Hospital length of stay | up to 90 days after start of intervention
Duration of renal replacement therapy | up to 28 days
Rate of renal replacement therapy | up to 28 days
Fluid balance | during intensive care unit stay
Dose of vasopressors | during intensive care unit stay
Duration of vasopressors | during hospital stay (up to 90 days after start of intervention)
Rate of infection during intensive care unit stay | during intensive care unit stay (up to 28 days after start of intervention)
Sequential organ failure assessment (SOFA) score | daily at days 1 to 14 after start of intervention
Sequential organ failure assessment (SOFA) score | daily at day 1 to 14, day 21 and day 28
Sequential organ failure assessment (SOFA) score | daily at days 28 after start of intervention
Need of renal replacement therapy (RRT) | 28 days after start of intervention
Need of renal replacement therapy (RRT) | 60 days after start of intervention
Need of renal replacement therapy (RRT) | 90 days after start of intervention
Need of renal replacement therapy (RRT) | 365 days after start of intervention
Rate of mortality | 90 days after start of intervention
Rate of mortality | 365 days after start of intervention
Rate of persistent renal dysfunction | 90 days after start of intervention
Rate of persistent renal dysfunction | 365 days after start of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Zarbock, MD, Study Chair — University Hospital Muenster, Dept. of Anesthesiology, Intensive Care Therapy and Pain Medicine
Locations (1):
- University Hospital Münster; 1Department of Anesthesiology, Intensive Care Medicine and Pain Medicine, Münster, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sadjadi M, Strauss C, von Groote T, Booke H, Schone LM, Sauermann L, Wempe C, Gerss J, Kellum J, Meersch M, Zarbock A. Effects of an extended therapeutic strategy versus standard-of-care therapy on persistent acute kidney injury in high-risk patients after major surgery: study protocol for the randomised controlled single-centre PrevProgAKI trial. BMJ Open. 2025 May 6;15(5):e097333. doi: 10.1136/bmjopen-2024-097333. PMID 40328648